CLINICAL TRIAL: NCT03597464
Title: A Randomized, Controlled, Double-blind, Continuation Study Comparing the Long-term Safety and Efficacy of Voclosporin (23.7 mg Twice Daily) With Placebo in Subjects With Lupus Nephritis
Brief Title: Aurinia Renal Assessments 2: Aurinia Renal Response in Lupus With Voclosporin
Acronym: AURORA 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aurinia Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AUR-VCS-2016-02
Record Dates: First submitted 2018-06-25; First posted 2018-07-24 (Actual); Results first posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-11

CONDITIONS: Lupus Nephritis
Keywords: lupus nephritis; calcineurin inhibitors; voclosporin
MeSH Terms: conditions — Lupus Nephritis | interventions — voclosporin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Voclosporin (Experimental): Voclosporin
  Interventions: Drug: Voclosporin
- Placebo Oral Capsule (Placebo Comparator): Placebo
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Voclosporin — Calcineurin inhibitor, oral, 23.7 mg twice daily (BID)
  Other Names: ISA247
  Arms: Voclosporin
Drug: Placebo Oral Capsule — Voclosporin placebo, oral, 3 capsules twice daily (BID)
  Arms: Placebo Oral Capsule

SUMMARY:
The purpose of this study is assess the long-term safety and tolerability of voclosporin compared with placebo for up to an additional 24 months following completion of treatment in the AURORA 1 study in subjects with lupus nephritis (LN).

DETAILED DESCRIPTION:
The aim of the Phase 3 continuation study (AURORA 2) is to assess the long-term safety and tolerability of voclosporin, added to the standard of care treatment in LN, for an additional 24 months, following a treatment period of 52 weeks in the AURORA 1 study (AUR-VCS-2016-01). All subjects will continue to receive background therapy of mycophenolate mofetil (MMF) and/or oral corticosteroids starting at the same dose as at the end of the AURORA 1 study. Subjects with LN, who have completed 52 weeks of treatment with study drug in the AURORA 1 study, will be eligible to enter the study. The long-term safety and tolerability of the drug combination will be assessed from its safety profile while demonstrating the continued ability to achieve and maintain long-term renal response.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have completed 52 weeks of treatment with study drug in the AURORA 1 study. Subjects who had a temporary interruption and successfully restarted study drug during the AURORA 1 study will be allowed with Medical Monitor approval.
2. Written informed consent before any study-specific procedures were performed.
3. In the opinion of the investigator, subject required continued immunosuppressive therapy.
4. Women of childbearing potential must continue to use effective contraception and have a negative urine pregnancy test at Month 12.
5. Subject is willing to continue taking oral mycophenolate mofetil (MMF) for the duration of the study.

Exclusion Criteria:

1. Currently taking or known need for any of the medications or food items listed in Section 7.8, Prohibited Therapy and Concomitant Treatment during the study.
2. Subjects currently requiring renal dialysis (hemodialysis or peritoneal dialysis) or expected to require dialysis during the study period.
3. A planned kidney transplant within study treatment period.
4. Subjects with any medical condition which, in the Investigator's judgment, may be associated with increased risk to the subject or may interfere with study assessments or outcomes.
5. Subjects who are pregnant, breast feeding or, if of childbearing potential, not using adequate contraceptive precautions.
6. Vaccines using live organisms, virus or bacterial, while taking the study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2019-09-29 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- AURORA Investigative Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rovin BH, Parikh SV, Hebert LA, Chan TM, Mok CC, Ginzler EM, Hooi LS, Brunetta P, Maciuca R, Solomons N. Lupus nephritis: induction therapy in severe lupus nephritis--should MMF be considered the drug of choice? Clin J Am Soc Nephrol. 2013 Jan;8(1):147-53. doi: 10.2215/CJN.03290412. Epub 2012 Aug 9. PMID 22879439
- [Background] Dooley MA, Jayne D, Ginzler EM, Isenberg D, Olsen NJ, Wofsy D, Eitner F, Appel GB, Contreras G, Lisk L, Solomons N; ALMS Group. Mycophenolate versus azathioprine as maintenance therapy for lupus nephritis. N Engl J Med. 2011 Nov 17;365(20):1886-95. doi: 10.1056/NEJMoa1014460. PMID 22087680
- [Background] Ling SY, Huizinga RB, Mayo PR, Larouche R, Freitag DG, Aspeslet LJ, Foster RT. Cytochrome P450 3A and P-glycoprotein drug-drug interactions with voclosporin. Br J Clin Pharmacol. 2014 Jun;77(6):1039-50. doi: 10.1111/bcp.12309. PMID 24330024
- [Background] Ling SY, Huizinga RB, Mayo PR, Freitag DG, Aspeslet LJ, Foster RT. Pharmacokinetics of voclosporin in renal impairment and hepatic impairment. J Clin Pharmacol. 2013 Dec;53(12):1303-12. doi: 10.1002/jcph.166. Epub 2013 Oct 8. PMID 23996158
- [Background] Mayo PR, Huizinga RB, Ling SY, Freitag DG, Aspeslet LJ, Foster RT. Voclosporin food effect and single oral ascending dose pharmacokinetic and pharmacodynamic studies in healthy human subjects. J Clin Pharmacol. 2013 Aug;53(8):819-26. doi: 10.1002/jcph.114. Epub 2013 Jun 4. PMID 23736966
- [Background] Busque S, Cantarovich M, Mulgaonkar S, Gaston R, Gaber AO, Mayo PR, Ling S, Huizinga RB, Meier-Kriesche HU; PROMISE Investigators. The PROMISE study: a phase 2b multicenter study of voclosporin (ISA247) versus tacrolimus in de novo kidney transplantation. Am J Transplant. 2011 Dec;11(12):2675-84. doi: 10.1111/j.1600-6143.2011.03763.x. Epub 2011 Sep 22. PMID 21943027
- [Derived] Avasare R, Drexler Y, Caster DJ, Mitrofanova A, Jefferson JA. Management of Lupus Nephritis: New Treatments and Updated Guidelines. Kidney360. 2023 Oct 1;4(10):1503-1511. doi: 10.34067/KID.0000000000000230. PMID 37528520

RESULTS

PARTICIPANT FLOW:
Groups:
- Voclosporin: Voclosporin 23.7 mg twice daily (BID) + Mycophenolate Mofetil + corticosteroid
- Placebo Oral Capsule: Placebo 23.7 mg twice daily (BID) + Mycophenolate Mofetil + corticosteroid
Period: Overall Study
Arm/Group | Voclosporin | Placebo Oral Capsule
Started | 116 | 100
Completed | 101 | 85
Not Completed | 15 | 15
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Lost to Follow-up | 3 | 1
Not completed — Pregnancy | 3 | 1
Not completed — Lack of Efficacy | 2 | 0
Not completed — Physician Decision | 2 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Adverse Event | 0 | 2
Not completed — Death | 0 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat is comprised of all subjects who were randomized treatment during AURORA 1 AND who consented to continue their treatment in AURORA 2. Baseline values were collected at the start of AURORA 1 but only for subjects that continued in AURORA 2. Intent-to-Treat population was used for analysis of all Outcome Measures. Safety population comprised all randomized subjects who took at least one dose of study treatment, and was used for AE and SAE reporting.
Groups:
- Voclosporin: Voclosporin 23.7 mg twice daily (BID) + Mycophenolate Mofetil (MMF) + corticosteroid
- Placebo Oral Capsule: Placebo 23.7 mg twice daily (BID) + Mycophenolate Mofetil (MMF) + corticosteroid
- Total: Total of all reporting groups
Arm/Group | Voclosporin | Placebo Oral Capsule | Total
Number analyzed (Participants) | 116 | 100 | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (10.31) | 35.4 (11.64) | 33.7 (11.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 88 | 193
  Male | 11 | 12 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 33 | 72
  Not Hispanic or Latino | 77 | 67 | 144
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 30 | 30 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 7 | 25
  White | 44 | 40 | 84
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 24 | 23 | 47
Region of Enrollment [Number; unit: participants] — Southeast Asia ("Asia Pacific") includes Japan, Malaysia, Philippines, Thailand, Taiwan & Vietnam.
  Europe ("Europe") includes Belarus, Croatia, Netherlands, Russia, Serbia, Spain, Turkey, Ukraine as well as South Africa.
  South America ("Latin America") includes Argentina, Brazil, Chile, Colombia, Dominican Republic, Guatemala, Mexico & Peru.
  participants
    United States | 15 | 9 | 24
    Southeast Asia | 29 | 27 | 56
    Europe | 38 | 37 | 75
    South America | 34 | 27 | 61
Lupus Nephritis (LN) history [Mean (Standard Deviation); unit: years] — Number of years since diagnosis of systemic lupus erythematosus (SLE), lupus nephritis (LN) and first significant proteinuria
  years
    Years since diagnosis of systemic lupus erythematosus (SLE) | 6.6 (6.66) | 7.3 (6.85) | 6.9 (6.75)
    Years since diagnosis of lupus nephritis (LN) | 4.8 (5.27) | 5.0 (5.23) | 4.9 (5.24)
    Years since first instance of significant proteinuria (>500 mg/day) | 5.0 (5.15) | 4.7 (4.49) | 4.8 (4.85)
Baseline Urine Protein Creatinine Ratio (UPCR) [Mean (Standard Deviation); unit: mg/mg] — Baseline Urine Protein Creatinine Ratio (UPCR) (Average of pre-randomisation values)
  mg/mg | 3.941 (2.5766) | 3.868 (2.4764) | 3.907 (2.5251)
Baseline estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73 m^2] — Baseline estimated Glomerular Filtration Rate Chronic Kidney Disease Epidemiology Collaboration (CKD-Epi formula) (lowest pre-randomisation value)
  mL/min/1.73 m^2 | 94.1 (31.36) | 92.0 (28.04) | 93.2 (29.82)

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events (AE) Profile and Routine Biochemical and Hematological Assessments.
Description: Number (and percent) of adverse events experienced during the AURORA 2 treatment period.
  To assess the long-term safety and tolerability of voclosporin compared with placebo for up to an additional 24 months following completion of treatment in the AURORA 1 study in subjects with LN.
Time Frame: Month 12 (AURORA 2 baseline) to Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | Voclosporin | Placebo Oral Capsule
Number analyzed (Participants) | 116 | 100
Participants
  Any treatment-emergent adverse event (TEAE) | 100 | 80
  Treatment-related TEAE | 28 | 21
  Serious TEAE | 21 | 23
  TEAE leading to study drug discontinuation | 11 | 17
  TEAE leading to death | 0 | 3
  Treatment-related TEAE leading to death | 0 | 0
  Disease-related TEAE | 50 | 34
  Disease-related serious TEAE | 7 | 11

2. Secondary Outcome: Number (and Percent) of Subjects in Renal Response
Description: Proportion of subjects in renal response defined as:
  * urine protein creatinine ratio (UPCR) of ≤0.5 mg/mg
  * estimated glomerular filtration rate (eGFR) ≥60 mL/min/1.73 m^2 or no confirmed decrease from baseline in eGFR of >20%
  * Received no rescue medication for LN
  * Did not receive more than 10 mg prednisone for ≥3 consecutive days or for ≥7 days in total during the 8 weeks prior to the renal response assessment.
Time Frame: Months 12 (AURORA 2 Baseline), 18, 24, 30 and 36
Measure: Count of Participants; unit: Participants
Arm/Group | Voclosporin | Placebo Oral Capsule
Number analyzed (Participants) | 116 | 100
Participants
  Renal Response - Month 12 | 61 | 34
  Renal Response - Month 18 | 74 | 46
  Renal Response - Month 24 | 65 | 43
  Renal Response - Month 30 | 69 | 42
  Renal Response - Month 36 | 59 | 39
Statistical Analysis 1: Comparison: Voclosporin vs Placebo Oral Capsule; Month 12 (AURORA 2 baseline); Test type: Other — The model is based on a logistic regression with terms for treatment, baseline UPCR, biopsy class, MMF use at baseline and region. Subjects who withdrew from the study prior to the visit assessments and thus provide insufficient visit data were defined as non-responders; p = 0.004, Regression, Logistic; Odds Ratio (OR) = 2.30, 95% CI 2-sided [1.30 to 4.05]
Statistical Analysis 2: Comparison: Voclosporin vs Placebo Oral Capsule; Month 18; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 2.19, 95% CI 2-sided [1.25 to 3.83]
Statistical Analysis 3: Comparison: Voclosporin vs Placebo Oral Capsule; Month 24; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.035, Regression, Logistic; Odds Ratio (OR) = 1.81, 95% CI 2-sided [1.04 to 3.16]
Statistical Analysis 4: Comparison: Voclosporin vs Placebo Oral Capsule; Month 30; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.005, Regression, Logistic; Odds Ratio (OR) = 2.24, 95% CI 2-sided [1.28 to 3.92]
Statistical Analysis 5: Comparison: Voclosporin vs Placebo Oral Capsule; Month 36; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.051, Regression, Logistic; Odds Ratio (OR) = 1.74, 95% CI 2-sided [1.00 to 3.03]

3. Secondary Outcome: Number (and Percent) of Subjects in Partial Renal Response
Description: Partial renal response defined as a 50% reduction from baseline in urine protein creatinine ratio (UPCR).
Time Frame: Months 12 (AURORA 2 baseline), 18, 24, 30 and 36
Measure: Count of Participants; unit: Participants
Arm/Group | Voclosporin | Placebo Oral Capsule
Number analyzed (Participants) | 116 | 100
Participants
  Partial Renal Response - Month 12 | 104 | 70
  Partial Renal Response - Month 18 | 96 | 68
  Partial Renal Response - Month 24 | 90 | 58
  Partial Renal Response - Month 30 | 85 | 61
  Partial Renal Response - Month 36 | 86 | 69
Statistical Analysis 1: Comparison: Voclosporin vs Placebo Oral Capsule; Month 12 (AURORA 2 baseline); Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.99, 95% CI 2-sided [1.88 to 8.46]
Statistical Analysis 2: Comparison: Voclosporin vs Placebo Oral Capsule; Month 18; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.008, Regression, Logistic; Odds Ratio (OR) = 2.50, 95% CI 2-sided [1.28 to 4.88]
Statistical Analysis 3: Comparison: Voclosporin vs Placebo Oral Capsule; Month 24; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 2.68, 95% CI 2-sided [1.46 to 4.91]
Statistical Analysis 4: Comparison: Voclosporin vs Placebo Oral Capsule; Month 30; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.040, Regression, Logistic; Odds Ratio (OR) = 1.86, 95% CI 2-sided [1.03 to 3.34]
Statistical Analysis 5: Comparison: Voclosporin vs Placebo Oral Capsule; Month 36; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.290, Regression, Logistic; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.75 to 2.58]

4. Secondary Outcome: Renal Flare as Adjudicated by the Clinical Endpoints Committee (CEC).
Description: A patient could experience a flare from the point they achieved a response (or recovery). Renal flares were judged according to the following criteria:
  * A reproducible increase to UPCR >1 mg/mg from a post-response baseline of <0.2 mg/mg or
  * an increase to UPCR >2 mg/mg from a post-response baseline between 0.2 to 1.0 mg/mg or
  * a doubling of UPCR for baseline values of UPCR >1 mg/mg
Time Frame: Month 12 (AURORA 2 baseline) to Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | Voclosporin | Placebo Oral Capsule
Number analyzed (Participants) | 116 | 100
Participants
  Subjects without adequate response or with flares | 39 | 46
  Subjects with adequate response and wothout flares | 77 | 54
Statistical Analysis 1: Comparison: Voclosporin vs Placebo Oral Capsule; Number of subjects with adequate renal response. This model is based on a logistic regression with terms for treatment, baseline urine protein creatinine ratio (UPCR), biopsy class, mycophenolate mofetil (MMF) use at baseline and region. An odds ratio < unity indicates benefit for voclosporin; Test type: Other; p = 0.045, Regression, Logistic; Odds Ratio (OR) = 0.56, 95% CI 2-sided [0.32 to 0.99]

5. Secondary Outcome: Change From AURORA 1 Baseline (i.e., Month 0) in Safety of Estrogens in Lupus Erythematosus National Assessment Systemic Lupus Erythematosus Disease Activity Index (SELENA-SLEDAI)
Description: Participants analyzed included all subjects who were randomized treatment during AURORA 1 AND who consented to continue their treatment in AURORA 2. Baseline values were collected at the start of AURORA 1 but only for those subjects that continued in AURORA 2.
  Assessment of Systemic Lupus Erythematosus (SLE) Disease Activity within the last 10 days. It scores 24 disease descriptors across 9 organ systems which are summed to a minimum of <2 (considered indicative of no activity) and maximum of 105 points. Scores are weighted and a score of 6 is considered clinically significant. Higher scores indicate worse disease activity.
Time Frame: Months 18, 24 and 36
Population: The number of subjects analyzed may not be aligned with overall number analyzed due to subjects withdrawing from study and missed study visits
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Voclosporin | Placebo Oral Capsule
Number analyzed (Participants) | 116 | 100
Scores on a scale
  Month 18: number analyzed (Participants) | 112 | 96
  Month 18 | -6.4 [-7.4 to -5.4] | -5.6 [-6.6 to -4.5]
  Month 24: number analyzed (Participants) | 100 | 84
  Month 24 | -6.8 [-7.7 to -5.9] | -6.1 [-7.0 to -5.1]
  Month 36: number analyzed (Participants) | 97 | 85
  Month 36 | -6.8 [-7.7 to -5.9] | -6.1 [-7.1 to -5.2]
Statistical Analysis 1: Comparison: Voclosporin vs Placebo Oral Capsule; Month 18; Test type: Superiority; p = 0.238, Mixed Models Analysis; Least Squares Mean difference = -0.8, 95% CI 2-sided [-2.1 to 0.5]
Statistical Analysis 2: Comparison: Voclosporin vs Placebo Oral Capsule; Month 24; Test type: Superiority; p = 0.215, Mixed Models Analysis; Least Squares Mean difference = -0.7, 95% CI 2-sided [-1.8 to 0.4]
Statistical Analysis 3: Comparison: Voclosporin vs Placebo Oral Capsule; Month 36; Test type: Superiority; p = 0.246, Mixed Models Analysis; Least Squares Mean difference = -0.7, 95% CI 2-sided [-1.8 to 0.5]

6. Secondary Outcome: Change From AURORA 1 Baseline (i.e., Month 0) in Urine Protein to Creatinine Ratio (UPCR)
Description: Participants analyzed included all subjects who were randomized treatment during AURORA 1 AND who consented to continue their treatment in AURORA 2. Baseline values were collected at the start of AURORA 1 but only for those subjects that continued in AURORA 2.
  Reductions in UPCR are indicative of better renal outcomes.
Time Frame: Months 12 (AURORA 2 baseline), 18, 24, 30 and 36
Population: The number of subjects analyzed may not be aligned with overall number analyzed due to early withdrawals from study and missed study visits
Measure: Least Squares Mean (Standard Error); unit: mg/mg
Arm/Group | Voclosporin | Placebo Oral Capsule
Number analyzed (Participants) | 116 | 100
mg/mg
  Month 12 (AURORA 2 baseline) | -3.17 (0.164) | -2.52 (0.175)
  Month 18: number analyzed (Participants) | 113 | 96
  Month 18 | -3.05 (0.216) | -2.42 (0.232)
  Month 24: number analyzed (Participants) | 105 | 81
  Month 24 | -3.18 (0.188) | -2.41 (0.202)
  Month 30: number analyzed (Participants) | 100 | 87
  Month 30 | -3.12 (0.219) | -2.21 (0.235)
  Month 36: number analyzed (Participants) | 99 | 87
  Month 36 | -3.00 (0.222) | -2.52 (0.236)
Statistical Analysis 1: Comparison: Voclosporin vs Placebo Oral Capsule; Month 12 (AURORA 2 baseline); Test type: Superiority; p = 0.001, Mixed Models Analysis; Least Squares Mean difference = -0.65, 95% CI 2-sided [-1.05 to -0.26]
Statistical Analysis 2: Comparison: Voclosporin vs Placebo Oral Capsule; Month 18; Test type: Superiority; p = 0.029, Mixed Models Analysis; Least Squares Mean difference = -0.63, 95% CI 2-sided [-1.20 to -0.07]
Statistical Analysis 3: Comparison: Voclosporin vs Placebo Oral Capsule; Month 24; Test type: Superiority; p = 0.002, Mixed Models Analysis; Least Squares Mean difference = -0.77, 95% CI 2-sided [-1.24 to -0.29]
Statistical Analysis 4: Comparison: Voclosporin vs Placebo Oral Capsule; Month 30; Test type: Superiority; p = 0.002, Mixed Models Analysis; Least Squares Mean difference = -0.91, 95% CI 2-sided [-1.49 to -0.33]
Statistical Analysis 5: Comparison: Voclosporin vs Placebo Oral Capsule; Month 36; Test type: Superiority; p = 0.106, Mixed Models Analysis; Least Squares Mean difference = -0.48, 95% CI 2-sided [-1.06 to -0.10]

7. Secondary Outcome: Change From AURORA 1 Baseline (i.e., Month 0) in Estimated Glomerular Filtration Rate (eGFR)
Description: Participants analyzed included all subjects who were randomized treatment during AURORA 1 AND who consented to continue their treatment in AURORA 2. Baseline values were collected at the start of AURORA 1 but only for those subjects that continued in AURORA 2.
  This endpoint incorporated Corrected eGFR values with a ceiling set to 90 mL/min/1.73 m^2
  Increases in eGFR levels are indicative of better renal outcomes.
Time Frame: Months 12 (AURORA 2 baseline), 18, 24, 30 and 36
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | Voclosporin | Placebo Oral Capsule
Number analyzed (Participants) | 116 | 100
mL/min/1.73 m^2
  Month 12 (AURORA 2 baseline) | 1.8 (1.08) | 4.4 (1.15)
  Month 18: number analyzed (Participants) | 114 | 96
  Month 18 | -0.2 (1.31) | 1.6 (1.40)
  Month 24: number analyzed (Participants) | 103 | 81
  Month 24 | -1.3 (1.48) | 0.9 (1.60)
  Month 30: number analyzed (Participants) | 99 | 85
  Month 30 | 0.2 (1.56) | -0.8 (1.67)
  Month 36: number analyzed (Participants) | 100 | 87
  Month 36 | -0.2 (1.69) | -2.0 (1.81)
Statistical Analysis 1: Comparison: Voclosporin vs Placebo Oral Capsule; Month 12 (AURORA 2 baseline); Test type: Superiority; p = 0.041, Mixed Models Analysis; Least Squares Mean difference = -2.7, 95% CI 2-sided [-5.3 to -0.1]
Statistical Analysis 2: Comparison: Voclosporin vs Placebo Oral Capsule; Month 18; Test type: Superiority; p = 0.292, Mixed Models Analysis; Least Squares Mean difference = -1.8, 95% CI 2-sided [-5.1 to 1.6]
Statistical Analysis 3: Comparison: Voclosporin vs Placebo Oral Capsule; Month 24; Test type: Superiority; p = 0.282, Mixed Models Analysis; Least Squares Mean difference = -2.2, 95% CI 2-sided [-6.1 to 1.8]
Statistical Analysis 4: Comparison: Voclosporin vs Placebo Oral Capsule; Month 30; Test type: Superiority; p = 0.659, Mixed Models Analysis; Least Squares Mean difference = 0.9, 95% CI 2-sided [-3.2 to 5.1]
Statistical Analysis 5: Comparison: Voclosporin vs Placebo Oral Capsule; Month 36; Test type: Superiority; p = 0.438, Mixed Models Analysis; Least Squares Mean difference = 1.8, 95% CI 2-sided [-2.8 to 6.4]

8. Secondary Outcome: Change From AURORA 1 Baseline (i.e., Month 0) in Urine Protein
Description: Participants analyzed included all subjects who were randomized treatment during AURORA 1 AND who consented to continue their treatment in AURORA 2. Baseline values were collected at the start of AURORA 1 but only for those subjects that continued in AURORA 2.
  Reductions in Urine Protein levels are indicative of better renal outcomes.
Time Frame: Months 12 (AURORA 2 baseline), 18, 24, 30 and 36
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Voclosporin | Placebo Oral Capsule
Number analyzed (Participants) | 116 | 100
mg/dL
  Month 12 (AURORA 2 baseline) | -302.4 (16.91) | -234.6 (18.05)
  Month 18: number analyzed (Participants) | 112 | 95
  Month 18 | -297.8 (23.41) | -210.1 (25.15)
  Month 24: number analyzed (Participants) | 104 | 81
  Month 24 | -295.8 (17.10) | -248.8 (18.51)
  Month 30: number analyzed (Participants) | 99 | 87
  Month 30 | -304.7 (19.23) | -231.6 (20.67)
  Month 36: number analyzed (Participants) | 99 | 86
  Month 36 | -280.7 (22.66) | -261.7 (24.01)
Statistical Analysis 1: Comparison: Voclosporin vs Placebo Oral Capsule; Month 12 (AURORA 2 baseline); Test type: Superiority; p = 0.002, Mixed Models Analysis; Least Squares Mean difference = -67.7, 95% CI 2-sided [-110.4 to -25.1]
Statistical Analysis 2: Comparison: Voclosporin vs Placebo Oral Capsule; Month 18; Test type: Superiority; p = 0.007, Mixed Models Analysis; Least Squares Mean difference = -87.7, 95% CI 2-sided [-151.2 to -24.2]
Statistical Analysis 3: Comparison: Voclosporin vs Placebo Oral Capsule; Month 24; Test type: Superiority; p = 0.035, Mixed Models Analysis; Least Squares Mean difference = -47.0, 95% CI 2-sided [-90.8 to -3.3]
Statistical Analysis 4: Comparison: Voclosporin vs Placebo Oral Capsule; Month 30; Test type: Superiority; p = 0.005, Mixed Models Analysis; Least Squares Mean difference = -73.1, 95% CI 2-sided [-123.5 to -22.6]
Statistical Analysis 5: Comparison: Voclosporin vs Placebo Oral Capsule; Month 36; Test type: Superiority; p = 0.537, Mixed Models Analysis; Least Squares Mean difference = -19.0, 95% CI 2-sided [-79.7 to 41.7]

9. Secondary Outcome: Change From AURORA 1 Baseline (i.e., Month 0) in Serum Creatinine (SCr)
Description: Participants analyzed included all subjects who were randomized treatment during AURORA 1 AND who consented to continue their treatment in AURORA 2. Baseline values were collected at the start of AURORA 1 but only for those subjects that continued in AURORA 2.
  Decreases in SCr levels can be indicative of better renal outcomes.
Time Frame: Months 12 (AURORA 2 baseline), 18, 24, 30 and 36
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Voclosporin | Placebo Oral Capsule
Number analyzed (Participants) | 116 | 100
mg/dL
  Month 12 (AURORA 2 baseline) | 0.051 (0.0207) | -0.034 (0.0221)
  Month 18: number analyzed (Participants) | 114 | 96
  Month 18 | 0.078 (0.0300) | 0.027 (0.0323)
  Month 24: number analyzed (Participants) | 103 | 81
  Month 24 | 0.117 (0.0429) | 0.060 (0.0466)
  Month 30: number analyzed (Participants) | 99 | 85
  Month 30 | 0.094 (0.0494) | 0.129 (0.0534)
  Month 36: number analyzed (Participants) | 100 | 87
  Month 36 | 0.119 (0.0597) | 0.197 (0.0644)
Statistical Analysis 1: Comparison: Voclosporin vs Placebo Oral Capsule; Month 12 (AURORA 2 baseline); Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Squares Mean difference = 0.084, 95% CI 2-sided [0.035 to 0.134]
Statistical Analysis 2: Comparison: Voclosporin vs Placebo Oral Capsule; Month 18; Test type: Superiority; p = 0.209, Mixed Models Analysis; Least Squares Mean difference = 0.051, 95% CI 2-sided [-0.029 to 0.131]
Statistical Analysis 3: Comparison: Voclosporin vs Placebo Oral Capsule; Month 24; Test type: Superiority; p = 0.353, Mixed Models Analysis; Least Squares Mean difference = 0.057, 95% CI 2-sided [-0.064 to 0.178]
Statistical Analysis 4: Comparison: Voclosporin vs Placebo Oral Capsule; Month 30; Test type: Superiority; p = 0.616, Mixed Models Analysis; Least Squares Mean difference = -0.036, 95% CI 2-sided [-0.176 to 0.105]
Statistical Analysis 5: Comparison: Voclosporin vs Placebo Oral Capsule; Month 36; Test type: Superiority; p = 0.372, Mixed Models Analysis; Least Squares Mean difference = -0.077, 95% CI 2-sided [-0.248 to 0.094]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) are events occurring from Month 12 of treatment (AURORA 2 baseline) up to 30 days after study treatment end in AURORA 2 (Month 37).
Description: Subjects are counted once within a system organ class and once for each unique preferred term.
Groups:
- Voclosporin: Voclosporin
  Voclosporin: Calcineurin inhibitor, oral, 23.7 mg BID
- Placebo Oral Capsule: Placebo
  Placebo Oral Capsule: Voclosporin placebo, oral, 3 capsules BID
Arm/Group | Voclosporin | Placebo Oral Capsule
All-Cause Mortality (participants affected / at risk) | 0/116 | 3/100
Serious Adverse Events (participants affected / at risk) | 21/116 | 23/100
Other Adverse Events (participants affected / at risk) | 84/116 | 60/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Voclosporin (N=116) | Placebo Oral Capsule (N=100)
Corona virus infection (Infections and infestations) | 2 (2) | 5 (5)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 2 (2)
Disseminated tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Lupus nephritis (Renal and urinary disorders) | 2 (2) | 3 (3)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (2) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 1 (1)
Malignant glaucoma (Eye disorders) | 0 (0) | 1 (1)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pericarditis lupus (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Voclosporin (N=116) | Placebo Oral Capsule (N=100)
Urinary tract infection (Infections and infestations) | 14 (22) | 8 (10)
Upper respiratory tract infection (Infections and infestations) | 10 (11) | 3 (6)
Viral upper respiratory tract infection (Infections and infestations) | 10 (10) | 4 (6)
Bronchitis (Infections and infestations) | 5 (5) | 4 (4)
Corona virus infection (Infections and infestations) | 5 (6) | 8 (9)
Gastroenteritis (Infections and infestations) | 5 (5) | 2 (2)
Herpes zoster (Infections and infestations) | 4 (4) | 7 (7)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 6 (8) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (4)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 5 (5) | 7 (9)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 10 (15) | 5 (5)
Nausea (Gastrointestinal disorders) | 3 (3) | 5 (6)
Lupus nephritis (Renal and urinary disorders) | 8 (9) | 1 (1)
Renal impairment (Renal and urinary disorders) | 4 (4) | 2 (2)
Proteinuria (Renal and urinary disorders) | 4 (6) | 1 (2)
Headache (Nervous system disorders) | 8 (12) | 5 (6)
Hypertension (Vascular disorders) | 10 (10) | 6 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Glomerular filtration rate decreased (Investigations) | 11 (14) | 5 (5)
Neutrophil count decreased (Investigations) | 2 (2) | 3 (3)
Oedema peripheral (General disorders) | 4 (4) | 8 (9)
Ligament sprain (Injury, poisoning and procedural complications) | 4 (5) | 1 (2)
Dry eye (Eye disorders) | 4 (4) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol: Protocol v1.0 (2017-10-13): https://cdn.clinicaltrials.gov/large-docs/64/NCT03597464/Prot_000.pdf
  • Study Protocol: Protocol v2.0 (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/64/NCT03597464/Prot_001.pdf
  • Study Protocol: Protocol v3.0 (2018-12-21): https://cdn.clinicaltrials.gov/large-docs/64/NCT03597464/Prot_002.pdf
  • Statistical Analysis Plan (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT03597464/SAP_003.pdf